CLINICAL TRIAL: NCT04319783
Title: Darolutamide + Consolidation Radiotherapy in Advanced Prostate Cancer Detected by PSMA
Acronym: DECREASE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Trans Tasman Radiation Oncology Group (Other)
Collaborators: Bayer (Industry); Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROG 19.06; U1111-1242-9233 (Other: UTN- World Health Organisation)
Record Dates: First submitted 2020-03-09; First posted 2020-03-24 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Advanced Prostate Carcinoma; Cancer of Prostate; PSA; Castrate Resistant Prostate Cancer
Keywords: Darolutamide; Consolidation Radiotherapy; PSA; PSMA PET; Prostate Cancer; Advanced Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Darolutamide (Experimental): Darolutimide 600mg BD
  Interventions: Drug: Darolutamide
- Local consolidation Radiotherapy + Darolutamide (Experimental): Darolutimide 600mg BD + local consolidative radiotherapy, with a biological equivalent dose of 30Gy/10fx or greater if delivered with SABR. SABR is the preferred treatment approach, however conventional radiotherapy is acceptable. To up to 5 sites of disease
  Interventions: Drug: Darolutamide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Darolutamide — Darolutamide alone
  Other Names: NUBEQA, Bayer HealthCare Pharmaceuticals Inc.
Radiation: Radiotherapy — Darolutamide + Consolidation Radiotherapy
  Arms: Local consolidation Radiotherapy + Darolutamide

SUMMARY:
Darolutamide is a drug that has a proven survival benefit in non-metastatic (M0) castrate resistant prostate cancer when using conventional imaging. However, it is estimated that >90% of patients have disease apparent when using PSMA PET. This study investigates the use of local consolidation radiotherapy in this cohort of men.

DETAILED DESCRIPTION:
This study explores the use of local consolidation therapy in the setting of Darolutamide in the initial diagnosis of metastatic castrate resistant prostate cancer (mCRPC). In the chemotherapy naïve mCRPC setting, the pattern of disease is of limited volume metastases (1-5) in 34%-40% of cases. As progression at known sites of macroscopic disease is the predominant cause of failure on systemic therapies, local consolidation therapy with stereotactic ablative body radiotherapy (SABR) may improve progression free survival (PFS) and overall survival (OS). This approach has been tested in the setting of lung cancer, in which consolidation SABR has resulted in OS benefit (HR of 0.40) in phase II studies. The novel approach of local consolidation therapy has not been tested as yet in mCRPC.

The secondary objective of this study proposal is to better understand the pattern of disease distribution at first diagnosis of CRPC. Previous studies have used conventional bone scan and CT imaging, and with these investigations the proportion of patients that are 'M0' is ~35%1. However, in the new era of PSMA PET, which is far more sensitive than conventional imaging, there exists a new group of men who are M0 on conventional imaging but are M1 on PSMA PET staging.

Thus, in the DECREASE study population, we expect the vast majority of patients with conventionally imaged 'M0 CRPC' will have disease detectable on PSMA PET scanning. In this context, the central hypothesis of this trial is that the addition of consolidation radiotherapy to darolutamide to PSMA detected sites of disease will improve the clinical outcome of patients compared to those patients receiving darolutamide alone.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age and provided written Informed Consent
* Histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Castration-resistant prostate cancer, defined as at least 2 consecutive PSA rises obtained at least 1 week apart in the setting of castrate testosterone levels
* Castrate level of serum testosterone (<1.7 nmol/l [50 ng/dl]) on gonadotrophin - releasing hormone (GnRH) agonist or antagonist therapy or after bilateral orchiectomy
* A baseline PSA level of at least 1ng per millilitre and a PSA doubling time of 10 months or less
* Adequate bone marrow reserve and organ function Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* At least 1 site of PSMA-avid disease on PSMA-PET/CT imaging in any of the following regions; At least 1 site of PSMA-avid disease on PSMA-PET/CT imaging in any of the following regions:

  * Local recurrence within the prostate gland or prostate bed
  * Regional lymph node disease (below the aortic bifurcation)
  * Extra-pelvic lymph node, bone or soft tissue metastatic disease

Exclusion Criteria:

* Patients with detectable metastases or a history of metastatic disease on conventional imaging
* Prior treatment with second-generation androgen receptor (AR) antagonists, CYP17 enzyme inhibitors or oral ketoconazole
* Use of oestrogens or 5-α reductase inhibitors or anti-androgens within 28 days before randomisation
* Use of systemic corticosteroid with a dose greater than the equivalent 10 mg of prednisone/day within 28 days before randomisation
* Radiotherapy within 12 weeks prior to randomisation
* Initiation of treatment with an osteoclast-targeted therapy to prevent skeletal-related events within 12 weeks before randomisation
* Any of the following within 6 months before randomisation: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft; congestive heart failure New York Heart Association (NYHA) Class III or IV
* Uncontrolled hypertension
* Prior malignancy
* Gastrointestinal disorder or procedure that expects to interfere significantly with the absorption of study treatment
* Unable to swallow study medications and comply with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Castration-resistant prostate cancer
Enrollment: 65 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Undetectable PSA at 12 months | 12 months
  Undetectable PSA at 12 months

SECONDARY OUTCOMES:
Radiological progression free survival | 36 months
  Radiological progression free survival
Distribution of disease on baseline PSMA-PET/CT imaging | 36 months
  Distribution of bone, nodal, visceral and recurrent primary disease on PSMA-PET/CT
Biochemical progression free survival | 36 months
  Biochemical progression free survival
Treatment related adverse event | 36 months
  Treatment related adverse events (CTCAE v 5.0)
Overall survival | 36 months
  Overall survival
Patterns of disease on PSMA PET/CT after 12 weeks of commencing Darolutamide, and at time of disease progression | 3 months
  PSMA avid disease at irradiated site / unirradiated site / bone / local / nodal / visceral

CONTACTS AND LOCATIONS:
Overall Officials: Shankar Siva, Study Chair — Peter MacCallum Cancer Centre, Australia; Arun Azad, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (16):
- Australia (15):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - GenesisCare Hurstville, Hurstville, New South Wales
  - GenesisCare North Shore, Saint Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital (ROPART), Raymond Terrace, Queensland
  - Princess Alexandra Hospital (ROPAIR), Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peter MacCallum Cancer Centre, Bendigo, Bendigo, Victoria
  - Peter MacCallum Cancer Centre, Box Hill, Box Hill, Victoria
  - Peter MacCallum Cancer Centre, Parkville, Melbourne, Victoria
  - Icon Cancer Centre Epworth, Richmond, Victoria
  - Western Health, St Albans, Victoria
  - GenesisCare Fiona Stanley Hospital, Murdoch, Western Australia
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No